CLINICAL TRIAL: NCT06996574
Title: A Pragmatic Randomised Prospective Multi-centre Non-inferiority Trial in Chronic Pain Patients With Closed-loop Spinal Cord Stimulation (CL-SCS) to Compare the Clinical Effectiveness and Cost Utility of an All-in-one Procedure With an At-home Screening Trial
Brief Title: Study to Compare the Clinical Effectiveness and Cost Utility of an All-in-one Procedure With an At-home Screening Trial
Acronym: All-in-one
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Professor Markus W Hollmann, Prof. dr. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024.1119
Record Dates: First submitted 2025-05-06; First posted 2025-05-30 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Neuromodulation; Chronic Pain Patients
Keywords: neuromodulation; chronic pain; SCS procedure; standard of care
MeSH Terms: conditions — Chronic Pain | interventions — Random Allocation

STUDY DESIGN:
Intervention Model Description: non inferiority
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- all-in-one (NTG) procedure (Experimental): all-in-one (NTG) procedure
  Interventions: Other: Randomization
- the established two-phase closed-loop SCS procedure with at-home screening trials (TG) (Placebo Comparator): Standard of Care
  Interventions: Other: Randomization

INTERVENTIONS:
Other: Randomization — The all-in-one (NTG) procedure versus the established two-phase closed-loop SCS procedure with at-home screening trials (TG) under everyday clinical practice, that can be used for clinical decision-making and to inform health policy decisions.

SUMMARY:
In 2019, the Dutch Healthcare Institute published a consensus report outlining when spinal cord stimulation (SCS) for chronic pain qualifies for reimbursement under Dutch health insurance. It mandates that adult patients with significant pain (VAS ≥50mm or NRS ≥5) undergo an at-home screening trial, which must show at least 50% pain reduction to proceed with permanent implantation. Screening trials give patients early access to the therapy, but they are expensive, often redundant, and pose risks such as infection. A recent UK study (TRIAL-STIM) found no significant difference in outcomes between patients who had screening trials and those who received an all-in-one SCS procedure, but the trial strategy incurred greater costs. Given these findings, and the fact that all-in-one procedures are already used in certain Dutch cases, it is reasonable to evaluate this approach more broadly. Therefore, a pragmatic, multi-centre, randomized non-inferiority trial will compare the effectiveness of the all-in-one procedure, no trial group (NTG) to the standard two-step approach, trial group (TG) in Dutch patients with chronic neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with chronic, neuropathic pain with an approved aetiology in the Netherlands PSPS (persistent spinal pain syndrome) PDN (painful diabetic neuropathy) CRPS (complex regional pain syndrome) SFN (small fibre neuropathy)
2. Suitable candidate according to the inclusion criteria of the Dutch "Standpoint on Neuromodulation in Chronic Pain" Adult patients ≥18 years Chronic pain ≥6 months Pain intensity of ≥50mm or ≥5 on VAS- or NRS-score respectively
3. Routinely selected for CL-SCS
4. Be willing to complete additional trial related questionnaires
5. Be willing and capable of giving informed consent.

Exclusion Criteria:

1. General exclusion criteria according to the Dutch "Standpoint on Neuromodulation in Chronic Pain":

   Drug abuse Pregnancy Coagulation disorder / Use of anticoagulation therapy which cannot be stopped temporarily Active infection Life expectation ≤12 months Intake questionnaires "PROMS neuromodulatie" not completed by the patient
2. Have an existing drug pump and/or SCS system or another active implantable device such as a pacemaker, deep brain stimulator (DBS), or sacral nerve stimulator (SNS)
3. Current or previous treatment with an implanted pain reduction device
4. Participation in another clinical trial that may confound the results of this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Pain Intensity on the Numeric Rating Scale (NRS) at 6 Months | up to 6 months post lead implant
  Pain intensity will be assessed using the 11-point Numeric Rating Scale (NRS), ranging from 0 (no pain) to 10 (worst imaginable pain). The primary outcome is the change in NRS score from baseline to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. dr. dr Hollmann W Prof. dr. dr., Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
We will describe the specific IPD that will be shared